CLINICAL TRIAL: NCT05149521
Title: A Consensus Study Using Nominal Group Technique to Develop Recommendations for a Comfort Intervention Package in Radiotherapy
Brief Title: Recommendations for a Radiotherapy Comfort Intervention Package Radiotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of the West of England (Other)
Collaborators: Somerset NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: HAS..21.10.024
Record Dates: First submitted 2021-09-23; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who have received radiotherapy: This is a consensus study with no interventions Patients who previously participated in COMFORT study interviews (NCT03984435)
  Interventions: Other: None - this is a consensus group study to develop an intervention
- Therapeutic radiographers who deliver radiotherapy: This is a consensus study with no interventions Therapeutic radiographers who previously participated in COMFORT study interviews (NCT03984435)
  Interventions: Other: None - this is a consensus group study to develop an intervention

INTERVENTIONS:
Other: None - this is a consensus group study to develop an intervention — None - this is a consensus group study to develop an intervention

SUMMARY:
A consensus study using nominal group technique is planned to develop recommendations for a comfort intervention package for radiotherapy with patients and therapeutic radiographers. This includes completed work from a systematic literature review (Prospero 59688) of comfort interventions applicable to radiotherapy and qualitative interviews (NCT03984435) with patients and therapeutic radiographers exploring comfort management in radiotherapy.

DETAILED DESCRIPTION:
Study Design

The aim of this study is to develop a radiotherapy comfort intervention package with patients and therapeutic radiographers.

The objectives are to:

Objective 1 - Identify and prioritise intervention components for inclusion in recommendations for a radiotherapy comfort intervention package.

Objective 2 - Determine the feasibility of delivering the component of the radiotherapy comfort intervention package.

Modified nominal group technique (NGT) will employed to develop recommendations for a comfort intervention package in radiotherapy in a consensus study with patients and therapeutic radiographers. This study follows earlier phases of the COMFORT study which included a systematic literature review of comfort interventions applicable to radiotherapy and qualitative interviews exploring comfort management in radiotherapy.

Study Participants

Patients

The inclusion criteria are: 1) diagnosed with a malignancy; 2) aged over 18 years owing to different treatment options for children and young adults; 3) recently referred for radiotherapy, currently receiving treatment or had had radiotherapy within the previous 3 months; 4) treatment delivery time exceeding 10 minutes (the time the patient is immobilised on the radiotherapy couch).

Therapeutic radiographers

The inclusion criteria are: 1) practicing radiographers; 2) administering radiotherapy with treatment delivery times exceeding 10 minutes per radiotherapy treatment session (the time the patient is immobilised on the radiotherapy couch).

The consensus study will be conducted by video conference.

Planned Size of Sample (if applicable)

6-12 participants (4-9 Patients and 2-3 Therapeutic radiographers)

Follow up duration (if applicable)

Follow up is not planned.

Planned Study Period

6 months

Research Question/Aim(s)

The aim of this study is to develop recommendations for a radiotherapy comfort intervention with patients and therapeutic radiographers.

ELIGIBILITY:
Inclusion Criteria:

Patients and therapeutic radiographers who previously participated in COMFORT study interviews

Exclusion Criteria:

Patients and therapeutic radiographers who did not participate in COMFORT study interviews

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Aiming to recruit between three main anatomical regions: head and neck, thorax and pelvis.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Prioritisation of comfort interventions applicable to radiotherapy | 1 month
  Consensus among patients and therapeutic radiographers using nominal group technique to achieve priority of comfort interventions

CONTACTS AND LOCATIONS:
Overall Officials: Simon Goldsworthy, MSc, Principal Investigator — Somerset NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Yes
The data will be the property of the Chief Investigator at the University of the West of England who is the data controller. Other researchers can request access to study data via the University of the West of England
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study completion for 10 years
Access Criteria: The data will be the property of the Chief Investigator at the University of the West of England who is the data controller.
  A full data management plan can be found in the UWE research repository at the following URL:
URL: https://uwe-repository.worktribe.com/

REFERENCES:
- [Background] Goldsworthy S, Palmer S, Latour JM, McNair H, Cramp M. A systematic review of effectiveness of interventions applicable to radiotherapy that are administered to improve patient comfort, increase patient compliance, and reduce patient distress or anxiety. Radiography (Lond). 2020 Nov;26(4):314-324. doi: 10.1016/j.radi.2020.03.002. Epub 2020 Mar 31. PMID 32245711